CLINICAL TRIAL: NCT06849934
Title: Reliability of Kinovea Software for Measurement of Transtibial Amputee Knee Angle During Walking
Brief Title: Reliability of Kinovea Software for Measurement of Transtibial Amputee Knee Kinematics
Status: Enrolling by invitation | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Şenay Çerezci Duygu, Asst. Prof., Saglik Bilimleri Universitesi
Other Study IDs: 2024-173
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-09

CONDITIONS: Amputee; Amputees
Keywords: amputee; motion analysis; kinematics; reliability

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary aim of this study was to find the reliability of Kinovea software in measuring parameters associated with sagittal plane knee kinematics during gait in transtibial amputees. The secondary objective was to calculate the absolute reliability by calculating the Standard Error of Measurement (SEM), SEM% and Minimal Detectable Change at 95% confidence interval (MDC95). The SEM value represents the extent to which a score changes during the repetition of the measurement. The MDC is the minimum change in the measurement that is considered a true change in the measured activity that is not due to error.

ELIGIBILITY:
Inclusion Criteria:

* Having a unilateral below-knee (transtibial) level amputation,
* Using a prosthesis and being able to walk with the prosthesis,
* Body mass index less than 30,
* No contracture in the intact or amputated knee.
* Not having had any surgery related to the knees.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have unilateral transtibial amputation
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Vİdeo Recording | From enrollment to the end of video record (10 minutes).
  The gait of the individuals will be recorded to determine the sagittal plane knee angular values during walking:
  Participants will be asked to wear comfortable clothing to avoid limitation of movement. Before recording any measurements, participants will be asked to walk a few laps around the test area to familiarize them with the procedure and the movements being measured. Video images of each participant will be acquired using a digital camera (Canon EOS600D) to capture the sagittal plane profile of the knee. The camera will be placed on a tripod at a height of 80 cm, 1.5 m away from the participants. The tripod will be placed on taped markers on the floor to maintain the same distance between the camera and the participants. All images will be transferred to a laptop and analyzed using Kinovea software, a free, open source software created for motion analysis (Kinovea, 0.8.15, http://www.kinovea.org/).

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Sciences, Ankara, Turkey (Türkiye)